CLINICAL TRIAL: NCT00196443
Title: Prospective, Randomized and Explorative Controlled Study About Influences of Compression Stockings on Skin's Barrier Function at Patients With Chronic Venous Insufficiency
Brief Title: The Influence of Compression Stockings on Skin's Barrier Function at Patients With Chronic Venous Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Bauerfeind AG, Zeulenroda, Germany (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bau-Phleb-17032005
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency

INTERVENTIONS:
Device: urea contained compressing stockings
Device: compressing stockings

SUMMARY:
The purpose of this study is to investigate if wearing of compression stockings influences the skin moisture. Conservative stockings are compared with urea containing compression stockings to find out if using urea prevents dehydration of the skin while wearing the urea compression stockings. Secondary aim was to find out if urea containing stockings increase the compliance to wear the compression stockings regulary by patients with diagnosed chronic venous insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Clincial diagnosis of chronic venous insufficiency
* Age: 18-80 years
* Patient's information and willingness to participate

Exclusion Criteria:

* Age under 18 years
* Lower limp edema not caused by venous insufficiency
* Acute deep venous thrombosis
* Arterial occlusive disease
* Diabetes mellitus with neuropathy or peripheral arterial disturbance of perfusion
* immobile Patients
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2005-06; Study Completion 2005-07

PRIMARY OUTCOMES:
skin moisture at day 0 and day 7
loss of water throughout epidermis at day 0 and day 7
throatiness of epidermis at day 0 and day 7

SECONDARY OUTCOMES:
compliance of patients at every day of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jünger, Prof. Dr., Principal Investigator — Clinic and Polyclinic of Dermatology, University of Greifswald; Andrea Ladwig, Study Chair — Clinic and Polyclinic of Dermatology, University of Greifswald
Locations (1):
- Clinic and Polyclinic of Dermatology, Ernst-Moritz-Arndt-University of Greifswald, Greifswald, Fleischmannstr. 42-44, Germany